CLINICAL TRIAL: NCT02552602
Title: The Role of Multivitamins in Pediatric HIV Management in Nigeria: A Randomized Controlled Study
Brief Title: The Role of Multivitamins in Pediatric HIV Management in Nigeria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Regina Esiovwa (Other)
Collaborators: University of the West of Scotland (Other); Brunel Healthcare Manufacturing Limited (Unknown); Partec Nigeria (Unknown); Panets Education Trust for Africa (PETA) (Unknown); Lagos State University (Other); Nigerian Institute of Medical Research (Other Government); Scottish Trace Element and Micronutrient Diagnostic and Research Laboratory, Glasgow (Unknown)
Responsible Party: Sponsor-Investigator, Regina Esiovwa, PhD Student, University of the West of Scotland
Organization: University of the West of Scotland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: REGPHD2015
Record Dates: First submitted 2015-09-09; First posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: HIV
Keywords: HIV; Multivitamins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Active Comparator): Study participants in this arm will be given Multivitamin A
  Interventions: Dietary Supplement: Multivitamin A
- Group B (Active Comparator): Study participants in this arm will be given Multivitamin B
  Interventions: Dietary Supplement: Multivitamin B
- Group C (Active Comparator): Study participants in this arm will be given Multivitamin C
  Interventions: Dietary Supplement: Multivitamin C

INTERVENTIONS:
Dietary Supplement: Multivitamin A — Multivitamin containing 7 micronutrients at recommended daily allowance (RDA)
  Arms: Group A
Dietary Supplement: Multivitamin B — Multivitamin containing 22 micronutrients at RDA
  Arms: Group B
Dietary Supplement: Multivitamin C — Multivitamin containing 22 micronutrients at three times the RDA
  Arms: Group C

SUMMARY:
Micronutrient deficiencies in people living with HIV have been reported. Multivitamins can address micronutrient deficiencies, however the benefits of multivitamins in people living with HIV is still debatable. While some multivitamin intervention studies have reported the benefits of multivitamins in HIV infection, some other studies have reported no statistical differences in outcomes of interest in intervention and control groups. With clear differences in composition and strength of the multivitamins used in the different studies, it is possible that some of the multivitamins used in some of the intervention studies may have been unable to meet existing micronutrient deficiencies. Hence there is a chance that higher strength multivitamins may be better able to correct these deficiencies and result in better outcomes. This study will therefore compare three different multivitamins varying in strength and composition to determine if any one of the three multivitamins will produce better health outcomes.

DETAILED DESCRIPTION:
The link between micronutrient deficiencies and advanced HIV disease has been reported. Micronutrient deficiencies in people living with HIV/AIDS (PLWHA) have been linked to reduced antioxidant levels and oxidative stress. In turn oxidative stress is believed to promote HIV disease progression. The use of multivitamins in PLWHA therefore has the potential to cut off the interconnections between micronutrient deficiencies and HIV disease progression. If beneficial, multivitamin use in PLWHA could result in improved health outcomes.

A number of studies have explored this possibility with different results. Differences in multivitamin strength and composition could have been responsible for the different results. Therefore, it is likely that increasing the strength and composition of the intervention multivitamin could possibly produce a single result of improved health outcomes across board. Hence this study will determine if multivitamins at higher strength can cause better health outcomes in study participants compared to lower strength multivitamins.

Multivitamin A is composed of 7 vitamins at recommended daily allowance (RDA), multivitamin B is made up of 22 micronutrients at RDA and multivitamin C is made up of 22 micronutrients at 3 times the RDA. These multivitamins were administered to the 190 study participants in a double blind randomized controlled study to determine if there would be any significant differences in health outcome of participants after 6 months of multivitamin use. All multivitamins regardless of their composition were manufactured to look identical and packaged in identical containers.

This double blind randomized controlled study is being conducted at the HIV treatment centers of the Nigerian Institute of Medical Research and the Lagos State University Teaching Hospital, both in Lagos Nigeria. At the design stage of the study, a feasibility study was carried out at both HIV treatment centers to assess the practicability and potential of success for this study. Following a successful feasibility study, ethical approval was applied for and obtained from each institution.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 5 - 12 years attending the outpatient clinic of the two HIV treatment centers who have tested positive to HIV
2. Children who can return for follow up during the 6 months of the study
3. Children with guardians who can give informed consent -

Exclusion Criteria:

1. Children enrolled in other studies
2. Guardians and children anticipating moving away from the study state
3. Children receiving immunosuppressive therapy

   -

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
CD4 count | 6 months
  A measure of immune competence. CD4 count could range from 500-1500 cells/mm3. Lower values can be seen with advancing HIV disease

SECONDARY OUTCOMES:
Serum selenium levels | 6 months
  To measure selenium deficiency. Range of 70µg/L -100µg/L have been proposed to describe adequacy of selenium levels in serum.
Serum zinc levels | 6 months
  To determine levels of zinc deficiency. 80µg/dL is often used as a cutoff point to signify deficiency in serum
Serum vitamin A levels | 6 months
  To determine vitamin A deficiency using cut off point of 0.7µmol/L for participants 5-6 years and 0.9µmol/L for participants 7-12 years
Red cell vitamin B6 levels | 6 months
  To identify B6 deficiency. 250-680 pmol/g haemoglobin will be the reference range used
Serum Copper levels | 6 months
  To evaluate copper deficiency. 12.5 to 22μmol/L will be the reference range used
Red cell manganese levels | 6 months
  To determine deficiency. Reference range not yet established
Red cell Magnesium | 6 months
  To determine deficiency levels. Reference range of 5.80-8.55 μmol/g haemoglobin will be used
Serum vitamin E levels | 6 months
  To determine deficiency. Reference range of 3.5 - 9.5 μmol/mmol cholesterol will be used
Red cell selenium levels | 6 months
  To measure selenium deficiency.3.6 - 10.6 nmol/g haemoglobin will be the reference range used
Red cell zinc levels | 6 months
  To determine zinc deficiency. 423-781 nmol/g haemoglobin will be the reference range used
Red cell Copper levels | 6 months
  To evaluate copper deficiency. 27.9-53.4 nmol/g haemoglobin will be the reference range used

OTHER OUTCOMES:
Hemoglobin (g/dl) | 6 months
  As part of routine tests
Serum Alanine aminotransferase (ALT) levels (U/L) | 6 months
  As part of routine tests
Serum Aspartate aminotransferase (AST) levels (IU/L) | 6 months
  As part of routine tests
Serum Bilirubin levels (mg/dl) | 6 months
  As part of routine tests
Serum Albumin levels (g/dl) | 6 months
  As part of routine tests
Serum Creatinine levels (mg/dl) | 6 months
  As part of routine tests
Serum Urea levels (mg/dl) | 6 months
  As part of routine tests
Serum C- Reactive Protein levels (mg/L) | 6 months
  As part of routine tests

CONTACTS AND LOCATIONS:
Overall Officials: Regina Esiovwa, Principal Investigator — University of the West of Scotland

REFERENCES:
- [Background] Akiibinu, M., Adeshiyan, A. and Olalekan, A. (2012) 'Micronutrients and markers of oxidative stress in symptomatic HIV positive/AIDS Nigerians: A call for adjuvant micronutrients therapy', The IIOAB Journal, 3, pp. 7-11.
- [Background] Baum MK, Campa A, Lai S, Sales Martinez S, Tsalaile L, Burns P, Farahani M, Li Y, van Widenfelt E, Page JB, Bussmann H, Fawzi WW, Moyo S, Makhema J, Thior I, Essex M, Marlink R. Effect of micronutrient supplementation on disease progression in asymptomatic, antiretroviral-naive, HIV-infected adults in Botswana: a randomized clinical trial. JAMA. 2013 Nov 27;310(20):2154-63. doi: 10.1001/jama.2013.280923. PMID 24281460
- [Background] Bhandari S, Banjara MR. Micronutrients Deficiency, a Hidden Hunger in Nepal: Prevalence, Causes, Consequences, and Solutions. Int Sch Res Notices. 2015 Jan 15;2015:276469. doi: 10.1155/2015/276469. eCollection 2015. PMID 27347513
- [Background] Bunupuradah T, Ubolyam S, Hansudewechakul R, Kosalaraksa P, Ngampiyaskul C, Kanjanavanit S, Wongsawat J, Luesomboon W, Pinyakorn S, Kerr S, Ananworanich J, Chomtho S, van der Lugt J, Luplertlop N, Ruxrungtham K, Puthanakit T; PREDICT study group. Correlation of selenium and zinc levels to antiretroviral treatment outcomes in Thai HIV-infected children without severe HIV symptoms. Eur J Clin Nutr. 2012 Aug;66(8):900-5. doi: 10.1038/ejcn.2012.57. Epub 2012 Jun 20. PMID 22713768
- [Background] Drain PK, Kupka R, Mugusi F, Fawzi WW. Micronutrients in HIV-positive persons receiving highly active antiretroviral therapy. Am J Clin Nutr. 2007 Feb;85(2):333-45. doi: 10.1093/ajcn/85.2.333. PMID 17284727
- [Background] Fawzi WW, Msamanga GI, Spiegelman D, Wei R, Kapiga S, Villamor E, Mwakagile D, Mugusi F, Hertzmark E, Essex M, Hunter DJ. A randomized trial of multivitamin supplements and HIV disease progression and mortality. N Engl J Med. 2004 Jul 1;351(1):23-32. doi: 10.1056/NEJMoa040541. PMID 15229304
- [Background] Guwatudde D, Wang M, Ezeamama AE, Bagenda D, Kyeyune R, Wamani H, Manabe YC, Fawzi WW. The effect of standard dose multivitamin supplementation on disease progression in HIV-infected adults initiating HAART: a randomized double blind placebo-controlled trial in Uganda. BMC Infect Dis. 2015 Aug 19;15:348. doi: 10.1186/s12879-015-1082-x. PMID 26285704
- [Background] Kaiser JD, Campa AM, Ondercin JP, Leoung GS, Pless RF, Baum MK. Micronutrient supplementation increases CD4 count in HIV-infected individuals on highly active antiretroviral therapy: a prospective, double-blinded, placebo-controlled trial. J Acquir Immune Defic Syndr. 2006 Aug 15;42(5):523-8. doi: 10.1097/01.qai.0000230529.25083.42. PMID 16868496
- [Background] Kupka R, Msamanga GI, Spiegelman D, Morris S, Mugusi F, Hunter DJ, Fawzi WW. Selenium status is associated with accelerated HIV disease progression among HIV-1-infected pregnant women in Tanzania. J Nutr. 2004 Oct;134(10):2556-60. doi: 10.1093/jn/134.10.2556. PMID 15465747
- [Background] Monteiro JP, Cruz ML, Mussi-Pinhata MM, Salomao RG, Jordao Junior A, Read JS, Pilotto JH, Cohen RA, Stoszek SK, Siberry GK. Vitamin A, vitamin E, iron and zinc status in a cohort of HIV-infected mothers and their uninfected infants. Rev Soc Bras Med Trop. 2014 Nov-Dec;47(6):692-700. doi: 10.1590/0037-8682-0226-2014. PMID 25626647
- [Background] Ndeezi G, Tylleskar T, Ndugwa CM, Tumwine JK. Effect of multiple micronutrient supplementation on survival of HIV-infected children in Uganda: a randomized, controlled trial. J Int AIDS Soc. 2010 Jun 3;13:18. doi: 10.1186/1758-2652-13-18. PMID 20525230
- [Background] Nkengfack GN, Torimiro JN, Englert H. Effects of antioxidants on CD4 and viral load in HIV-infected women in sub-Saharan Africa - dietary supplements vs. local diet. Int J Vitam Nutr Res. 2012 Feb;82(1):63-72. doi: 10.1024/0300-9831/a000095. PMID 22811378
- [Background] Pugliese C, Patin RV, Palchetti CZ, Claudio CC, Gouvea Ade F, Succi RC, Amancio OM, Cozzolino SM, Oliveira FL. Assessment of antioxidants status and superoxide dismutase activity in HIV-infected children. Braz J Infect Dis. 2014 Sep-Oct;18(5):481-6. doi: 10.1016/j.bjid.2014.02.003. Epub 2014 Apr 26. PMID 24780364
- [Background] Semba RD, Tang AM. Micronutrients and the pathogenesis of human immunodeficiency virus infection. Br J Nutr. 1999 Mar;81(3):181-9. doi: 10.1017/s0007114599000379. PMID 10434844
- [Background] Semeere AS, Nakanjako D, Ddungu H, Kambugu A, Manabe YC, Colebunders R. Sub-optimal vitamin B-12 levels among ART-naive HIV-positive individuals in an urban cohort in Uganda. PLoS One. 2012;7(7):e40072. doi: 10.1371/journal.pone.0040072. Epub 2012 Jul 2. PMID 22768330
- [Background] Sharma B. Oxidative stress in HIV patients receiving antiretroviral therapy. Curr HIV Res. 2014;12(1):13-21. doi: 10.2174/1570162x12666140402100959. PMID 24694264
- [Background] Shin DH, Martinez SS, Parsons M, Jayaweera DT, Campa A, Baum MK. Relationship of Oxidative Stress with HIV Disease Progression in HIV/HCV Co-infected and HIV Mono-infected Adults in Miami. Int J Biosci Biochem Bioinforma. 2012;2(3):217-223. doi: 10.7763/ijbbb.2012.v2.104. PMID 23504530
- [Background] Shivakoti R, Christian P, Yang WT, Gupte N, Mwelase N, Kanyama C, Pillay S, Samaneka W, Santos B, Poongulali S, Tripathy S, Riviere C, Berendes S, Lama JR, Cardoso SW, Sugandhavesa P, Tang AM, Semba RD, Campbell TB, Gupta A; NWCS 319 and PEARLS Study Team. Prevalence and risk factors of micronutrient deficiencies pre- and post-antiretroviral therapy (ART) among a diverse multicountry cohort of HIV-infected adults. Clin Nutr. 2016 Feb;35(1):183-189. doi: 10.1016/j.clnu.2015.02.002. Epub 2015 Feb 10. PMID 25703452
- [Background] Singh G, Pai RS. Dawn of antioxidants and immune modulators to stop HIV-progression and boost the immune system in HIV/AIDS patients: An updated comprehensive and critical review. Pharmacol Rep. 2015 Jun;67(3):600-5. doi: 10.1016/j.pharep.2014.12.007. Epub 2014 Dec 24. PMID 25933975
- [Background] UNICEF (2006) Preventing and controlling micronutrient deficiencies in populations affected by an emergency. Available at: http://www.unicef.org/nutrition/files/Joint_Statement_Micronutrients_March_2006.pdf (Accessed: 5 September 2015).
- [Background] Visser ME, Maartens G, Kossew G, Hussey GD. Plasma vitamin A and zinc levels in HIV-infected adults in Cape Town, South Africa. Br J Nutr. 2003 Apr;89(4):475-82. doi: 10.1079/BJN2002806. PMID 12654165
- [Derived] Esiovwa R, Rankin J, David A, Disu E, Wapmuk A, Amoo O. The Role of Multimicronutrient Supplementation in Pediatric HIV Management in Nigeria: A Randomized Controlled Study. J Pediatric Infect Dis Soc. 2021 Mar 26;10(2):112-117. doi: 10.1093/jpids/piaa025. PMID 32202619